CLINICAL TRIAL: NCT00460304
Title: The Effect of Pramlintide on Meal Time Insulin Bolus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Care Center (Industry)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-01
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Type 1 Diabetes
Keywords: Type I diabetes; Insulin pump; Continuous glucose monitoring; Insulin to carbohydrate ratio; Correction factor; Pramlintide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pramlintide
Procedure: continuous glucose monitoring

SUMMARY:
The primary objective is to establish the mean percentage of change in the insulin-to-carbohydrate ratio due to pramlintide treatment once a maximum tolerated dose or 6 mcg before each meal is reached. The secondary objective is to establish which insulin bolus wave form is associated with the lowest post-bolus without hypoglycemia in subjects treated with maximum pramlintide dosage.

DETAILED DESCRIPTION:
Pramlintide. an amylinomimetic, is effective in reducing post-meal glucose by non-insulin means. As such, when patients requiring insulin treatment are treated with pramlintide, the bolus insulin does must be reduced. Current recommendations suggest a 50% reduction but in our experience and that of a recent study this appears excessive. By using continuous glucose monitoring(CGM) to guide pre-meal insulin treatment, we will determine the percentage reduction in meal time insulin bolus comparing pre-pramlintide to maximum pramlintide treatment. We anticipate that the reduction in bolus dosage will be about 25%. In addition, the secondary aim of this study is to determine which bolus pattern, standard, square or dual wave, provides the best post-meal glucose control with pramlintide therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: >17
* Type I diabetes
* Onset of diabetes >3 months
* Use of insulin pump >3 months
* Hb A1C <8.9%
* Demonstrated compliance to clinic visits
* Demonstrated knowledge and use of bolus dosing calculations, carbohydrate counting, use of insulin pump and blood glucose meter
* Monitor blood glucose >4/day

Exclusion Criteria:

* Pregnancy or nursing
* Recent (within last 3 months) factor that may cause change in insulin sensitivity, e.g. severe emotional or physical stress, recent significant infection or surgery. etc.
* Renal failure (creatinine >1.5 mg/dl
* Symptomatic gastroparesis
* Using a medication that would interfere with insulin sensitivity
* Treatment with extenatide or DPP IV inhibitor within the last 4 weeks
* HbA1C change >0.9 % within the last 3 months
* Significant change in eating or activity pattern
* Weight change of >1.9 kg within the last 3 months
* ALT >3 times upper limits of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The mean ICR from Vist 3a-e and 4a-e will be compared. Percentage reduction of ICR will be calculated. From these the mean ICR will be calculated. | 12-10-07

SECONDARY OUTCOMES:
The mean post-meal glucose from the four hour period after beginning a meal will be averaged for each bolus wave form. Then the three wave form mean glucose results will be compared. | 12-10-07

CONTACTS AND LOCATIONS:
Overall Officials: Allen B King, MD, Principal Investigator — Diabetes Care Center; Gary S Wolfe, RN, CCM, Study Director — Diabetes Care Center

REFERENCES:
- [Background] Edelman S, Garg S, Frias J, Maggs D, Wang Y, Zhang B, Strobel S, Lutz K, Kolterman O. A double-blind, placebo-controlled trial assessing pramlintide treatment in the setting of intensive insulin therapy in type 1 diabetes. Diabetes Care. 2006 Oct;29(10):2189-95. doi: 10.2337/dc06-0042. PMID 17003291
- [Background] Symlin (package insert) San Diego, CA Amylin Pharmacetucials. 2005
- [Background] King AB, Armstrong DU. Basal bolus dosing: a clinical experience. Curr Diabetes Rev. 2005 May;1(2):215-20. doi: 10.2174/1573399054022794. PMID 18220597
- [Background] King AB, Armstrong DU. A prospective evaluation of insulin dosing recommendations in patients with type 1 diabetes at near normal glucose control: Basal dosing. J Diabetes Sci Technol. 2007 Jan;1(1):36-41. doi: 10.1177/193229680700100106. PMID 19888377
- [Background] King AB, Armstrong DU. A prospective evaluation of insulin dosing recommendations in patients with type 1 diabetes at near normal glucose control: bolus dosing. J Diabetes Sci Technol. 2007 Jan;1(1):42-6. doi: 10.1177/193229680700100107. PMID 19888378
- [Background] Young AA, Gedulin B, Vine W, Percy A, Rink TJ. Gastric emptying is accelerated in diabetic BB rats and is slowed by subcutaneous injections of amylin. Diabetologia. 1995 Jun;38(6):642-8. doi: 10.1007/BF00401833. PMID 7672483
- [Background] Gedulin BR, Rink TJ, Young AA. Dose-response for glucagonostatic effect of amylin in rats. Metabolism. 1997 Jan;46(1):67-70. doi: 10.1016/s0026-0495(97)90170-0. PMID 9005972
- [Background] Rushing PA, Lutz TA, Seeley RJ, Woods SC. Amylin and insulin interact to reduce food intake in rats. Horm Metab Res. 2000 Feb;32(2):62-5. doi: 10.1055/s-2007-978590. PMID 10741687
- [Background] Gross TM, Mastrototaro JJ. Efficacy and reliability of the continuous glucose monitoring system. Diabetes Technol Ther. 2000;2 Suppl 1:S19-26. doi: 10.1089/15209150050214087. No abstract available. PMID 11469628